CLINICAL TRIAL: NCT01675518
Title: A Phase 1 Randomized, Double-blind, Placebo-controlled, Dose-escalation Study to Assess the Safety, Tolerability, Pharmacokinetics (PK) and Pharmacodynamics (PD) of a Single Oral Administration of ASP7991 in Healthy Volunteers
Brief Title: A Study to Assess the Safety, Pharmacological Effect and Plasma Concentration of ASP7991 After Single Oral Administration to Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple
Other Study IDs: 7991-CL-0001
Record Dates: First submitted 2012-08-28; First posted 2012-08-30 (Estimated); Last update posted 2012-08-30 (Estimated); Status verified 2012-08

CONDITIONS: Healthy; Pharmacokinetics of ASP7991
Keywords: Plasma concentration; ASP7991; food effect; PTH (parathyroid hormone)
MeSH Terms: interventions — ASP7991

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (9):
- Part-1 dose 1 (Experimental)
  Interventions: Drug: ASP7991
- Part-1 dose 2 (Experimental)
  Interventions: Drug: ASP7991
- Part-1 dose 3 (Experimental)
  Interventions: Drug: ASP7991
- Part-1 dose 4 (Experimental)
  Interventions: Drug: ASP7991
- Part-1 dose 5 (Experimental)
  Interventions: Drug: ASP7991
- Part-1 dose 6 (Experimental)
  Interventions: Drug: ASP7991
- Part-1 placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- Part-2 fed (Experimental)
  Interventions: Drug: ASP7991
- Part-2 fasted (Experimental)
  Interventions: Drug: ASP7991

INTERVENTIONS:
Drug: ASP7991 — oral
  Arms: Part-1 dose 1; Part-1 dose 2; Part-1 dose 3; Part-1 dose 4; Part-1 dose 5; Part-1 dose 6; Part-2 fasted; Part-2 fed
Drug: Placebo — oral
  Arms: Part-1 placebo

SUMMARY:
This study is to assess the safety, tolerability, plasma concentration and pharmacodynamics of ASP7991 after single oral administration to healthy volunteers. In part-1, ASP7991 is administered in a dose escalation design. In part-2, plasma concentration changes of ASP7991 in fasted and fed conditions are compared.

DETAILED DESCRIPTION:
This study consists of two parts. In Part 1, the study will begin as a single rising dose escalation design under randomized double-blind and fasting conditions. In each dose group, volunteers will be randomized to receive an oral administration of either active drug (ASP7991) or placebo. The dose escalation will be determined after blinded safety assessment.

Part 2 is a study to evaluate the effect of food intake. ASP7991 will be administered to volunteers under 2 conditions, fasting and fed, on 2-way crossover method.

ELIGIBILITY:
Inclusion Criteria:

* Healthy, as judged by the investigator/sub investigator based on the results of physical examination obtained before study drug administration
* Body weight: ≥50.0 kg, <80.0 kg
* BMI: ≥17.6, <26.4
* Serum corrected calcium concentration: ≥9.0mg/dL, <10.4 mg/dL

Exclusion Criteria:

* Received any investigational drugs in other clinical or post-marketing studies within 120 days before screening
* Donated 400 mL of whole blood within 90 days, 200 mL of whole blood within 30 days, or blood components within 14 days before screening
* Received medication (including marketed drug) within 7 days before hospitalization, vitamin preparation including vitamin D and supplement including calcium or is scheduled to receive medication
* A deviation from normal criteria range of 12-lead ECG (QT evaluation)
* A deviation from the normal range in clinical laboratory tests
* Highly sensitive cardiac troponin T (at screening): ≥0.014 ng/mL
* History of drug allergies
* Upper gastrointestinal disease (e.g. nausea, vomiting, stomachache) within 7 days before admission
* Concurrent or previous hepatic disease (e.g., viral hepatitis, drug-induced liver injury)
* Concurrent or previous endocrine disorders (e.g.,hyperthyroidism, aberration in growth hormone)

Ages: 20 Years to 44 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2012-01; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
The safety of ASP7991 assessed by the incidence of adverse events, vital signs, laboratory tests, 12-lead ECGs and Holter ECGs | for 96 hours after dosing

SECONDARY OUTCOMES:
Plasma Concentration of unchanged drug :Cmax, tmax, AUClast, AUCinf, t1/2, CL/F | for 96 hours after dosing
  Blood samples are collected at the following times: redose and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12,16, 24, 48, 72 and 96 hours
Urinary concentrations of unchanged drug: Aelast，Aelast%, CLr | for 96 hour after dosing
  Urine samples are collected at the following times: redose and 0-4, 4-8, 8-12, 12-24, 24-36, 36-48, 48-72, 72-96 hours
plasma parathyroid hormon concentration | for 96 hours after dosing
  Blood samples are collected at the following times: redose and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12,16, 24, 48, 72 and 96 hours

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Astellas Pharma Inc
Locations (1):
- Kantou, Japan